CLINICAL TRIAL: NCT00488735
Title: Subacute and Chronic, Non-specific Back and Neck Pain: Cognitive-behavioral Rehabilitation Compared With Traditional Primary Care Concerning Sick-listing and Health-care Visits. A Randomized Controlled Trial, 18-month Follow-up
Brief Title: Subacute and Chronic, Non-specific Back and Neck Pain: Cognitive-behavioral Rehabilitation vs. Traditional Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KarolinskaI
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2007-06

CONDITIONS: Back Pain; Neck Pain
Keywords: Randomized controlled trial; Back pain; Neck pain; Rehabilitation; Cognitive-behavioral; Primary care; Sick-listing; Health-care utilization.
MeSH Terms: conditions — Back Pain; Neck Pain; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive-behavioral rehabilitation
Behavioral: Traditional primary care

SUMMARY:
BACKGROUND

Non-specific back and neck pain (BNP) dominates sick-listing. A program of cognitive-behavioral rehabilitation for subacute and chronic BNP was compared, with 18-month follow-up, with traditional primary care concerning sick-listing and health-care visits.

METHODS

After stratification to age (44 (years) and younger/45 and older) and subacute/chronic BNP (= full-time sick-listed 43-84/85-730 days respectively), 125 primary-care patients were randomized to a rehabilitation center or continued health-center care. Outcome measures were Return-to-work (=the proportion who regained work ability for at least 30 consecutive days), the proportion with Work ability at different time points, Total sick-listing (expressed in whole days) and the total number of Visits (to physicians, physiotherapists etc.) 1-18 months and corresponding six-month periods. For the analyses were used t-test, z-test, generalized estimating equations and a mixed, linear model.

DETAILED DESCRIPTION:
Numbers within parenthesis refers to the place of order in the citation list and within brackets in the link list below.

B A C K G R O U N D

In Sweden, as all over the industrial world, unspecific back and neck pain (BNP) dominates sick-listing (1). Primary care is the appropriate source of treatment of most patients with BNP (2). However, the Swedish traditional primary care lacks the capacity of such an assignment [1]. While the number of practicing physicians is in line with OECD standards, Sweden has, relatively seen, few physicians within primary care. Our overall aim was to compare a program of cognitive-behavioral-rehabilitation at a rehabilitation center for patients with subacute and chronic BNP with traditional primary care. The specific aim of this study was to answer the question: Will the outcome, with an 18-month follow-up, differ concerning sick-listing and number of health-care visits?

M E T H O D S

PARTICIPANTS: One-hundred-and-twenty-five patients were recruited by 42 family doctors at 12 health centers.

INCLUSION AND EXCLUSION CRITERIA: See below

INTERVENTIONS: Cognitive-behavioral rehabilitation: The medical, biomechanical and psychosocial obstacles to working were mapped out. A physiotherapist let the patient into graded activity (3). A behaviorist offered cognitive-behavioral therapy. A health adviser taught applied relaxation (4). A physician prescribed medicine when needed. Then the individual management was replaced by team conferences. A rehabilitation plan was drawn up. The patient gradually returned to work. The end of rehabilitation came when the final aim was achieved or when it was clear that work ability would not be attained. Participation in the rehabilitation group did not exclude the patient from seeking other care also.

Traditional primary care: The hub of Swedish primary care is the health centres. Besides family doctors, their staff consists of, among others, physiotherapists and social workers. In total, the health centers of this study engaged 84 family doctors and served a population of 148 000 individuals, i.e. slightly less than 0.6, as compared with an OECD-average of 0.8, family doctors/1000 population [2]. Participation in the health-center group excluded the patient from turning to the rehabilitation center but not from any other health-care, for example, orthopedist consultation.

DATA COLLECTION: Sick-listing data were provided by the Stockholm County Social Insurance Agency. Data of the treatment at the rehabilitation center were collected from its medical journals. As to the rest, health-care data were obtained from follow-up forms.

OUTCOME MEASURES: See below.

POWER CALCULATION: It originated from a retrospective preliminary study of 172 patients at the rehabilitation centre and from a forecast of the probability of ever regaining work ability for patients with full-time sick-listing for back pain in traditional care (5). The proportion of patients with any degree of work ability at the end of the rehabilitation was 76% and, for the patients with subacute and chronic BNP, 89% and 73% respectively. The average probability of regaining work ability in the case of continued management within traditional care was calculated for each one of the 172 patients according to their period of sick-listing at the start of the rehabilitation and was on average 49% as to be compared with the 76% who really regained work ability. The smallest difference that we wished to demonstrate was 22%. With a significance level of .05 and a power of 80% 154 patients had to be included, and to allow a certain dropout, 170 patients.

PREMATURE STOP OF RECRUITMENT: The recruitment was discontinued in January 2004 at 125 patients. The reason was that in April 2004 a large back-rehabilitation centre started in a neighboring municipality. We presumed that many of the planned future patients of the health-center group would be referred to that centre and get a management that could no longer be defined as traditional primary care.

INCLUSION PROCEDURE: A patient who fulfilled the criteria and agreed to participate was interviewed by telephone by a research assistant. The patients who still qualified saw the assistant at the health center and went through a start form. Then the assistant carried out a 10-test package, including a lift test. The reliability of that test procedure was confirmed in a separate study (6). Then the randomization was made with stratifications to age 44 and younger and 45 and older, and to subacute BNP and chronic BNP, i.e. full-time sick listed 43-84 and 85-730 days respectively. The stratifications were made out from the results of the preliminary study. Randomization envelopes were used. The patients of the rehabilitation group started the program at the centre within one week. The patients of the health-center group continued at their health-centers (= traditional primary care).

FOLLOW-UP: Six, 12 and 18 months after inclusion, the patients were sent follow-up forms.

ANALYSES AND STATISTICS: A p-value<.05 was considered statistically significant. For interval data were used t-test, ordinal data Wilcoxon rank-sum test and proportions z-test. Total sick-listing as well as Visits for the pre- and post-inclusion six-months periods was compared with a mixed-linear model (7).

ELIGIBILITY:
Inclusion Criteria:

1. Working age up to and including 59 years.
2. Sick-listed full-time for BNP for at least 42 days and at most 730 days.
3. Able to manage tolerably well to fill in forms.

Exclusion Criteria:

1. Temporary disability pension or disability pension being paid or in preparation.
2. A primary need of action by a hospital specialist.
3. Pregnancy and diseases which would probably make rehabilitation impracticable (for example, advanced pulmonary disease).
4. Whiplash-associated disorders as a primary obstacle to working.
5. Previous rehabilitation at the rehabilitation centre.
6. Other multidisciplinary rehabilitation going on or planned.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2000-08; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Return-to-work=the proportion of patients who during 1-18 months regained a degree of work ability>0 for at least 30 days in succession. | 18 months.

SECONDARY OUTCOMES:
Work ability (=the proportion with work ability>0). Total sick-listing=the sum of sick-listing of any degree, expressed in whole days. Visits=the total number of consultations to different health-care staff, for example, physicians or physiotherapists. | Work ability: 18 months. Total sick-listing: 36 months (18 months preceding and after inclusion). Visits: 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Erik Strender, Professor, Study Chair — Centre for Family Medicine, Karolinska Institutet
Locations (1):
- Centre for Family Medicine, Stockholm, Huddinge, Sweden

REFERENCES:
- [Background] Alexanderson K, Norlund A. Swedish Council on Technology Assessment in Health Care (SBU). Chapter 1. Aim, background, key concepts, regulations, and current statistics. Scand J Public Health Suppl. 2004;63:12-30. doi: 10.1080/14034950410021808. No abstract available. PMID 15513650
- [Background] Söderström M, Englund L: Treatment of neck and low back pain in primary care. In Neck and back pain. The scientific evidence of causes, diagnosis, and treatment. Edited by Nachemson A, Jonson E. Philadelphia: Lippincott, Williams & Williams; 2000:383-398.
- [Background] Lindstrom I, Ohlund C, Eek C, Wallin L, Peterson LE, Fordyce WE, Nachemson AL. The effect of graded activity on patients with subacute low back pain: a randomized prospective clinical study with an operant-conditioning behavioral approach. Phys Ther. 1992 Apr;72(4):279-90; discussion 291-3. doi: 10.1093/ptj/72.4.279. PMID 1533941
- [Background] Linton SJ: Utility of cognitive-behavioral psychological treatments. In Neck and back pain. The scientific evidence of causes, diagnosis, and treatment. Edited by Nachemson A, Jonson E. Philadelphia: Lippincott, Williams & Williams; 2000:361-381.
- [Background] Waddell G. Low back pain: a twentieth century health care enigma. Spine (Phila Pa 1976). 1996 Dec 15;21(24):2820-5. doi: 10.1097/00007632-199612150-00002. PMID 9112705
- [Background] Brown H, Prescott R: Applied mixed models in medicine. Edinburgh: John Wiley & Sons LTD; 199-259, 2001.
- [Result] Lindell O, Eriksson L, Strender LE. The reliability of a 10-test package for patients with prolonged back and neck pain: could an examiner without formal medical education be used without loss of quality? A methodological study. BMC Musculoskelet Disord. 2007 Apr 3;8:31. doi: 10.1186/1471-2474-8-31. PMID 17407580
- [Derived] Lindell O, Johansson SE, Strender LE. Predictors of stable return-to-work in non-acute, non-specific spinal pain: low total prior sick-listing, high self prediction and young age. A two-year prospective cohort study. BMC Fam Pract. 2010 Jul 20;11:53. doi: 10.1186/1471-2296-11-53. PMID 20646286
- [Derived] Lindell O, Johansson SE, Strender LE. Subacute and chronic, non-specific back and neck pain: cognitive-behavioural rehabilitation versus primary care. A randomized controlled trial. BMC Musculoskelet Disord. 2008 Dec 30;9:172. doi: 10.1186/1471-2474-9-172. PMID 19116007